CLINICAL TRIAL: NCT00358176
Title: A Multicenter, Double-blind, Randomized, Active-controlled, Parallel Group, Noninferiority Study Comparing 75mg Risedronate Dosed on 2 Consecutive Days Monthly With 5mg Daily Risedronate in the Treatment of Postmenopausal Osteoporosis as Assessed Over 24 Months.
Brief Title: Risedronate 75mg Dosed on 2 Consecutive Days Monthly in the Treatment of Osteoporosis in Postmenopausal Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Procter and Gamble (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC6063; HMR4003M/3001
Record Dates: First submitted 2006-07-28; First posted 2006-07-31 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2009-12

CONDITIONS: Osteoporosis Postmenopausal
Keywords: Treatment osteoporosis postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Risedronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Risedronate (HMR4003)

SUMMARY:
To confirm the non-inferiority of 75 mg risedronate tablets taken on 2 consecutive days per month as compared to 5 mg risedronate tablets taken daily in increasing bone mass in lumbar spine in postmenopausal women with osteoporosis.

To confirm the efficacy of 75 mg risedronate tablets taken on 2 consecutive days per month in postmenopausal women with osteoporosis in increasing bone mass in proximal femur, femoral neck and femoral trochanter and decreasing bone resorption.

To confirm general safety of 75 mg risedronate tablets taken on 2 consecutive days per month as compared to 5 mg risedronate taken daily.

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting all of the following criteria were considered for enrollment into the study :

·Ambulatory, healthy postmenopausal women with :

* Natural menopause and more than 5 years after their last menstrual period.
* Or surgical menopause and more than 5 years after surgery (blood hormone tests required for subjects less than 65 years of age who had uterus removed without removal of ovaries at time of surgery).

Osteoporosis (lumbar spine T-score more than 2.5 SD below the mean value in normal young women or more than 2.0 SD below the mean value in normal young women and at least 1 fracture of a vertebra (thoracic-lumbar T4-L4)).

Exclusion Criteria:

Subjects with any of the following criteria were not considered for enrollment into the study :

·Women who have received hormone replacement therapy (with estrogen by mouth and/or progestogen and/or androgen) or raloxifene, or other bone active drugs, such as calcitonin, calcitriol/calcidiol/alfacalcidol, parathyroid hormone or any bisphosphonate within 3 months before first dose of study medication.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1231 (Actual)
Dates: Start 2004-07; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in lumbar spine bone mineral density (BMD) at
Month 12 measured by dual-energy X-ray absorptiometry (DXA).

SECONDARY OUTCOMES:
Efficacy:Percent change from baseline in Lumbar spine BMD at times other than Month 12, Proximal femur BMD and Bone turnover markers.
Safety: AEs, clinical laboratory values, bone biopsies.
Intact serum parathyroid hormone (PTH 1-84)before treatment and after 3, 12 and 24 months of treatment in approximately 25% of randomly selected trial participants.
Physical examination before treatment and after 12 and 24 months of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (11):
- Sanofi-Aventis, Bridgewater, New Jersey, United States
- Sanofi-Aventis, San Isidro, Argentina
- Sanofi-Aventis, Macquarie Park, Australia
- Sanofi-Aventis, Laval, Canada
- Sanofi-Aventis, Prague, Czechia
- Sanofi-Aventis, Paris, France
- Sanofi-Aventis, Beirut, Lebanon
- Sanofi-Aventis, Warsaw, Poland
- Sanofi-Aventis, Midrand, South Africa
- Sanofi-Aventis, Istanbul, Turkey (Türkiye)
- Sanofi-Aventis, Guildford Surrey, United Kingdom